CLINICAL TRIAL: NCT03568045
Title: Feasibility Pilot of Bright Light in the Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 2000022284; 1K23HL138229-01A1 (NIH); 1R03HL157009-01 (NIH)
Record Dates: First submitted 2018-06-05; First posted 2018-06-26 (Actual); Results first posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Circadian Rhythm Sleep Disorder, Unspecified
Keywords: circadian misalignment; entrainment; zeitgeber; bright light; critical illness
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Critical Illness

STUDY DESIGN:
Intervention Model Description: a pilot randomized control trial of 3 cohort groups.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Usual care, standard light (Active Comparator): Patients will be enrolled within 30 hours of noon on enrollment day (e.g. at or after 6am on the prior calendar day). Enrollment will occur before noon, and the day of enrollment is termed study day 1.
  Patients will undergo monitoring (light levels, circadian alignment), but otherwise have usual care.
  Interventions: Device: standard light
- 10,000 lux bright light, 4 hours (Experimental): Patients will be enrolled within 30 hours of noon on enrollment day (e.g. at or after 6am on the prior calendar day). Enrollment will occur before noon, and the day of enrollment is termed study day 1.
  Patients will undergo monitoring (light levels, circadian alignment), starting on study day 1. Patients will be exposed to bright light from 8am to noon starting on study day 2 and continuing through study day 5. Bright light exposure will occur in the Intensive Care Unit (ICU) and on the floor if the patient is transferred.
  Feasibility metrics will be collected.
  Interventions: Device: 10,000 lux bright light, 4 hours
- 10,000 lux bright light, 8 hours (Experimental): Patients will be enrolled within 30 hours of noon on enrollment day (e.g. at or after 6am on the prior calendar day). Enrollment will occur before noon, and the day of enrollment is termed study day 1.
  Patients will undergo monitoring (light levels, circadian alignment), starting on study day 1. Patients will be exposed to bright light from 8am to 4pm starting on study day 2 and continuing through study day 5. Bright light exposure will occur in the Intensive Care Unit (ICU) and on the floor if the patient is transferred.
  Feasibility metrics will be collected.
  Interventions: Device: 10,000 lux bright light, 8 hours

INTERVENTIONS:
Device: standard light — usual care
  Arms: Usual care, standard light
Device: 10,000 lux bright light, 4 hours — Bright light will be delivered by a free-standing 10,000 lux device that will be positioned next to the patient's head of bed. At the estimated distance of 36 inches from light source to the patient, we anticipate approximately a 1,250 lux dose at the patient's eye. Light will be delivered from 8am to noon.
  Other Names: Bright light, 4 hours
  Arms: 10,000 lux bright light, 4 hours
Device: 10,000 lux bright light, 8 hours — Bright light will be delivered by a free-standing 10,000 lux device that will be positioned next to the patient's head of bed. At the estimated distance of 36 inches from light source to the patient, we anticipate approximately a 1,250 lux dose at the patient's eye. Light will be delivered from 8am to 4pm.
  Other Names: Bright light, 8 hours
  Arms: 10,000 lux bright light, 8 hours

SUMMARY:
To evaluate the feasibility of providing daytime bright light in the ICU in a pilot randomized controlled trial.

DETAILED DESCRIPTION:
To evaluate the feasibility of providing daytime bright light in the ICU in a pilot randomized controlled trial. Feasibility will be assessed via the following metrics: daytime bright light is acceptable and tolerable to patients and has high fidelity and sustainability as an intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Hospital admission ≤30 hours at noon on enrollment day
2. Expected to say in the Medical Intensive Care Unit ≥24 hours after enrollment
3. Age ≥50 years
4. History of hypertension based on chart review and presence of 1 or more home blood pressure medications
5. Able to understand English

Exclusion Criteria:

1. At significant risk for pre-existing circadian abnormalities:

   * Severe chronic brain injury (Injury greater than 30 days ago resulting in the inability to live independently) OR Acute brain injury of any severity (Injury less than 30 days ago including acute intracranial bleed, traumatic brain injury, central nervous system infection, tumor)
   * Documented circadian disorder (<1% population) or blind/disease of the optic nerve
   * Current history of substance abuse including alcohol (use in last 30 days)
   * Current or recent (last 1 year) shiftwork
2. Home medications include: melatonin, melatonin agonist
3. Transferred from an outside hospital, long-term care, rehabilitation, or acute care facility
4. History of bipolar disease (Bright light therapy possibly unsafe in this population).
5. Paralyzed (due to injury, disease or medications)
6. Diagnosed with hepatic encephalopathy in the setting of end-stage liver disease
7. Homeless

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Knauert, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, York Street Campus, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care, Standard Light: Patients will be enrolled within 30 hours of noon on enrollment day (e.g. at or after 6am on the prior calendar day). Enrollment will occur before noon, and the day of enrollment is termed study day 1.
  Patients will undergo monitoring (light levels, circadian alignment), but otherwise have usual care.
  standard light: usual care
- 10,000 Lux Bright Light, 4 Hours: Patients will be enrolled within 30 hours of noon on enrollment day (e.g. at or after 6am on the prior calendar day). Enrollment will occur before noon, and the day of enrollment is termed study day 1.
  Patients will undergo monitoring (light levels, circadian alignment), starting on study day 1. Patients will be exposed to bright light from 8am to noon starting on study day 2 and continuing through study day 5. Bright light exposure will occur in the Intensive Care Unit (ICU) and on the floor if the patient is transferred.
  Feasibility metrics will be collected.
  10,000 lux bright light, 4 hours: Bright light will be delivered by a free-standing 10,000 lux device that will be positioned next to the patient's head of bed. At the estimated distance of 36 inches from light source to the patient, we anticipate approximately a 1,250 lux dose at the patient's eye. Light will be delivered from 8am to noon.
- 10,000 Lux Bright Light, 8 Hours: Patients will be enrolled within 30 hours of noon on enrollment day (e.g. at or after 6am on the prior calendar day). Enrollment will occur before noon, and the day of enrollment is termed study day 1.
  Patients will undergo monitoring (light levels, circadian alignment), starting on study day 1. Patients will be exposed to bright light from 8am to 4pm starting on study day 2 and continuing through study day 5. Bright light exposure will occur in the Intensive Care Unit (ICU) and on the floor if the patient is transferred.
  Feasibility metrics will be collected.
  10,000 lux bright light, 8 hours: Bright light will be delivered by a free-standing 10,000 lux device that will be positioned next to the patient's head of bed. At the estimated distance of 36 inches from light source to the patient, we anticipate approximately a 1,250 lux dose at the patient's eye. Light will be delivered from 8am to 4pm.
Period: Overall Study
Arm/Group | Usual Care, Standard Light | 10,000 Lux Bright Light, 4 Hours | 10,000 Lux Bright Light, 8 Hours
Started | 2 | 9 | 5
Completed | 2 | 9 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All consented and enrolled patients included in baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care, Standard Light | 10,000 Lux Bright Light, 4 Hours | 10,000 Lux Bright Light, 8 Hours | Total
Number analyzed (Participants) | 2 | 9 | 5 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (5.7) | 73.6 (10.6) | 73.6 (11.9) | 72.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 8
  Male | 1 | 6 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 8 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 2 | 7 | 5 | 14
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Tolerance (Time): Percent of Intended Treatment Hours That Patient Continues With the Delivery of Bright Light
Description: Percent of intended treatment hours that patient continues with the delivery of bright light once exposed to bright light.
Time Frame: Study Day 2-5
Population: Enrolled patients who were randomized to either bright light treatment arm.
Measure: Mean (Standard Error); unit: percentage of intended treatment hours
Arm/Group | Usual Care, Standard Light | 10,000 Lux Bright Light, 4 Hours | 10,000 Lux Bright Light, 8 Hours
Number analyzed (Participants) | 0 | 9 | 5
percentage of intended treatment hours |  | 59 (11) | 61 (13)

2. Secondary Outcome: Acceptance: Percent of Patients/Surrogates Who Agree to Bright Light When Initially Described
Description: Percent of patients/surrogates who agree to study enrollment including bright light when initially described to them.
Time Frame: Study Day 1 (enrollment)
Population: Eligible patients who were approached for consent.
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Patients: Eligible patients who were approached for consent.
Arm/Group | Eligible Patients
Number analyzed (Participants) | 67
Participants | 59

3. Secondary Outcome: Tolerance (Symptoms): Percent of Patients Who Develop Eye Strain, Headache or Visual Disturbance.
Description: Percent of patients who develop eye strain, headache or visual disturbance.
Time Frame: Study Day 2-5
Population: All enrolled patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care, Standard Light | 10,000 Lux Bright Light, 4 Hours | 10,000 Lux Bright Light, 8 Hours
Number analyzed (Participants) | 2 | 9 | 5
Participants | 0 | 2 | 1

4. Secondary Outcome: Fidelity: Percent of Time Per Day That Device Delivers the Planned Dose of Light
Description: Percent of time per day that device delivers the planned dose of light (out of 4 or 8 hours depending on intervention arm).
Time Frame: Study Day 2-5
Population: Enrolled patients randomized to either bright light treatment arm.
Measure: Mean (Standard Error); unit: percentage of time per day
Arm/Group | Usual Care, Standard Light | 10,000 Lux Bright Light, 4 Hours | 10,000 Lux Bright Light, 8 Hours
Number analyzed (Participants) | 0 | 9 | 5
percentage of time per day |  | 55 (8) | 55 (11)

5. Secondary Outcome: Sustainability: Percent of Intended Intervention Days That the Device is Used.
Description: Percent of intended intervention days that the device is used. For this metric, days that the patient refuses bright light will not be included in "intended intervention days."
Time Frame: Study Day 2-5
Population: Enrolled patients randomized to either bright light treatment arm.
Measure: Mean (Standard Error); unit: percentage of intervention days used
Arm/Group | Usual Care, Standard Light | 10,000 Lux Bright Light, 4 Hours | 10,000 Lux Bright Light, 8 Hours
Number analyzed (Participants) | 0 | 9 | 5
percentage of intervention days used |  | 94 (6) | 88 (7)

ADVERSE EVENTS:
Time Frame: Patients were followed for outcomes until discharge from the index MICU/hospital admission, up to study day 5.
Arm/Group | Usual Care, Standard Light | 10,000 Lux Bright Light, 4 Hours | 10,000 Lux Bright Light, 8 Hours
All-Cause Mortality (participants affected / at risk) | 1/2 | 2/9 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/2 | 2/9 | 0/5
Other Adverse Events (participants affected / at risk) | 0/2 | 2/9 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care, Standard Light (N=2) | 10,000 Lux Bright Light, 4 Hours (N=9) | 10,000 Lux Bright Light, 8 Hours (N=5)
Death (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) — Death during index hospitalization.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care, Standard Light (N=2) | 10,000 Lux Bright Light, 4 Hours (N=9) | 10,000 Lux Bright Light, 8 Hours (N=5)
Visual strain (Eye disorders) | 0 (0) | 2 (2) | 0 (0) — Visual strain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT03568045/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT03568045/ICF_001.pdf